CLINICAL TRIAL: NCT04313569
Title: Arthroscopic Versus Conservative Treatment of Degenerative Meniscal Tear in Middle Aged Patients in Regard to Pain & Knee Function: Comparative Study
Brief Title: Arthroscopic Versus Conservative Treatment of Degenerative Meniscal Tear in Middle Aged Patients in Regard to Pain & Knee Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan9
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Knee Pain Chronic
Keywords: Degenerative meniscal tear; arthroscopic partial meniscectomy; conservative treatment; medial meniscal tear

STUDY DESIGN:
Intervention Model Description: Arthroscopic meniscectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (No Intervention): Use of medications, like analgesic, muscle relaxants, non-steroidal anti-inflammatory drugs (NSAID) and local painkillers, depending on the patient condition, and physiotherapy, lifestyle and daily activity modification, patient education about positioning of the knee
- Arthroscopic menisctomy (Other)
  Interventions: Procedure: Arthroscopic menisctomy

INTERVENTIONS:
Procedure: Arthroscopic menisctomy — Arthroscopic medial menisctomy
  Arms: Arthroscopic menisctomy

SUMMARY:
The study is prospective comparative study, conducted in Erbil teaching hospital on 60 patients, their age ranging between 40 and 60 years. All were clinically diagnosed to have degenerative medial meniscal tear then confirmed by MRI. Thirty patients were treated conservatively, thirty patients were treated arthroscopically.

ELIGIBILITY:
Inclusion Criteria:

1. Atraumatic continuous pain in medial aspect of knee affecting daily activities, for more than one month despite the treatment of general physician.
2. Grade 3 degenerative tear of medial meniscus approved on MRI.

Exclusion Criteria:

1. Meniscal tear due to trauma.
2. Any rheumatologic knee disease.
3. MRI showing ligament injury, loose bodies, tumors and osteochondral defects.
4. Former surgery of knee and lower limb fractures in the last year.
5. Knee joints with osteoarthritis graded 2 or more according to Kellgren-Lawrence scale (Kellgren and Lawrence, 1957) on weight-bearing knee x-ray.
6. Lateral meniscus tear.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Lysholm Knee Scoring Scale | All patients were reviewed and evaluated one year, by Lysholm score
  Lysholm Knee score scale has (8) parts (swelling, pain, squatting, support, stair climbing, limping, locking and instability). Score of 100 means no problems in knee.
Visual analogue score | All patients were reviewed and evaluated one year, by Visual Analogue score scales
  Ten points Visual Analogue Score scale used in order to meassure the severity of knee pain during the study. Zero meaning no pain while 10 meaning the most severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Sherwan Hamawandi, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No